CLINICAL TRIAL: NCT02326987
Title: A Randomized, Open, Single-dose, 3-treatment, 3-period, 6-sequence Crossover Study in Healthy Male Subjects to Evaluate the Pharmacokinetics of GLA5PR GLARS-NF1 Tablet 150mg and LYRICA® Capsule 75mg
Brief Title: A Clinical Trial to Compare The Pharmacokinetics of A Pregabalin GLARS-NF1 Tablet 150mg With Immediate Release Formulation and to Assess The Effect of High Fat Diet in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GLA5PR-103
Record Dates: First submitted 2014-12-10; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GLA5PR GLARS-NF1 tab.150mg(fasted) (Experimental): GLA5PR GLARS-NF1 tab. 150mg/day(Pregabalin 150mg once a day)
  Interventions: Drug: Pregabalin 150mg
- GLA5PR GLARS-NF1 tab.150mg(after high fat meal) (Experimental): GLA5PR GLARS-NF1 tab. 150mg/day(Pregabalin 150mg once a day)
  Interventions: Drug: Pregabalin 150mg
- Lyrica Capsule 75mg(after high fat meal) (Active Comparator): Lyrica Capsule 150mg/day(Pregabalin 75mg twice a day)
  Interventions: Drug: Pregabalin 75mg

INTERVENTIONS:
Drug: Pregabalin 150mg — GLA5PR GLARS-NF1 tablet 150mg/day(Pregabalin 150mg once a day)
  Other Names: GLA5PR GLARS-NF1 tab.150mg
  Arms: GLA5PR GLARS-NF1 tab.150mg(after high fat meal); GLA5PR GLARS-NF1 tab.150mg(fasted)
Drug: Pregabalin 75mg — Lyrica Capsule 150mg/day(Pregabalin 75mg twice a day)
  Other Names: Lyrica Capsule 75mg
  Arms: Lyrica Capsule 75mg(after high fat meal)

SUMMARY:
The purpose of this clinical trial is to compare the pharmacokinetic characteristics of GLA5PR GLARS tablet 150mg and Lyrica Capsule 75mg.

GLA5PR GLARS tablet 150mg is a New Formulation which is made by GL Pharm Tech.

GLARS(Geometrically Long Absorption Regulated System) is New Solution to Sustained Absorption by Extending the Absorption Site.

To overcome the shortcomings of the currently existing sustained release drug delivery technologies the investigators have recently developed a novel drug delivery system to enable a drug to be dissolved irrespective of the surrounding environment and further absorbed up to colon. The investigators coined this "Geometrically Long Absorption Regulated System(GLARS)".

DETAILED DESCRIPTION:
Basically, this system is a triple-layered tablet, comprised of upper and lower layers that swell and draw a sufficient amount of water, plus a highly water - soluble middle layer that rapidly draw water into the tablet core simultaneously.

The water drawn into the tablet (about 3 to 4 times the weight of the tablet itself) functions as an additional media which enables additional and later drug release out of the dosage form. This serves to overcome the shortage of surrounding media that has been reported to be one of the key reasons for mal-absorption of a drug in colon.

As the middle layer induces a rapid water draw into the tablet core, the penetrated water also diffuses to the upper and lower layers, which makes the tablet to rapidly swell and controls drug release.

At virtually the same time, the swollen upper and lower layers form to surround a lateral side of the middle layer, which can, in turn, further control drug release.

This relatively rigid swollen matrix structure makes drug release not affected by surrounding mechanical flux, which can provide relatively consistent in vivo drug release irrespective of degree of gastrointestinal motility.

ELIGIBILITY:
Inclusion Criteria:

* 20~45 years old, Healthy Adult Male Subject
* 17.5~30.5kg/m2(BMI) and ≥ 45kg

Exclusion Criteria:

* SBP ≥ 140mmHg or DBP ≥ 90mmHg

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
AUClast | 36hrs
  Pharmacokinetic of Pregabalin
Cmax | 36hrs
  Pharmacokinetic of Pregabalin

SECONDARY OUTCOMES:
AUCinf | 36hrs
  Pharmacokinetic of Pregabalin
Tmax | 36hrs
  Pharmacokinetic of Pregabalin
t1/2 | 36hrs
  Pharmacokinetic of Pregabalin
CL/F | 36hrs
  Pharmacokinetic of Pregabalin
Vd/F | 36hrs
  Pharmacokinetic of Pregabalin

REFERENCES:
- [Derived] Kim TE, Jeon JY, Gu N, Chang Kwon M, Kim MG. Comparative Pharmacokinetics of a Controlled-release Pregabalin Tablet (GLA5PR GLARS-NF1) and an Immediate-release Pregabalin Capsule in Healthy Male Volunteers. Clin Ther. 2018 Dec;40(12):2112-2124. doi: 10.1016/j.clinthera.2018.10.017. Epub 2018 Nov 27. PMID 30497798